CLINICAL TRIAL: NCT04044157
Title: Non-invasive Cardiac Output Monitoring in Children During the Perioperative Period - a Pilot Study
Brief Title: Cardiac Output in Children During Anesthesia
Acronym: COC
Status: Completed | Type: Observational
Sponsor: Laszlo Vutskits (Other)
Responsible Party: Sponsor-Investigator, Laszlo Vutskits, Head of Pediatric Anesthesia, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: BASEC 2019-00884
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Perioperative Period; Cardiac Output; Pediatric Anesthesia; Arterial Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-invasive measurement of cardiac output — cardiac output will be non-invasivaly measured by means of electrical cardiometry
  Other Names: no other intervention

SUMMARY:
This study investigates cardiac output in young children under 18 months of age during the perioperative period by means of electrical cardiometry.

DETAILED DESCRIPTION:
Young children are particularly prone to hemodynamic instability during the perioperative period which, in turn, may lead to organ morbidity. Currently, in routine surgical procedures in otherwise healthy children, hemodynamic status in the perioperative period is primarily assessed by non-invasive systemic blood pressure management. While this approach can detect systemic arterial hypotension, it does not provide us with guidance on whether the decrease in blood pressure is the result of changes in cardiac output and/or in systemic vascular resistance. This information would be important to know since treatment modalities may differ.

Recent technical development in electrical cardiometry allows us to non-invasively monitor cardiac output. The accuracy of the method has been validated in neonatal and pediatric cohorts, and electrical cardiometry is now regularly used to monitor cardiac output in the perioperative setting. Nevertheless, the temporal patterns of cardiac output changes in otherwise healthy young children undergoing routine surgical procedures have not been systematically reported. This information is important since it will increase our understanding of hemodynamic changes in small children during anesthesia/surgery and would ultimately lead to a better anesthesia care in this patient population.

The primary objective of this pilot exploratory observational study is to describe temporal patterns of cardiac output in young children ( under18 months of age) during the perioperative period. The secondary objectives are to describe how changes in cardiac output are associated with (i) non-invasively-measured systemic arterial blood pressure; (ii) near-infrared spectroscopy; (iii) other anesthesia factors (arterial oxygen saturation, concentration of anesthesia agents, CO2 levels).

ELIGIBILITY:
Inclusion Criteria:

* age 0 to 17 months included
* undergo general anesthesia for surgery that is expected to last more than 30 minutes (combines anesthesia and surgical time)
* parental/guardian permission (informed consent) obtained
* ASA 1-3 status

Exclusion Criteria:

* structural/anatomical anomaly or other circumstances (e.g. patient positioning) making it difficult to apply the sensors to the body
* history of congenital heart diseases
* known allergy to electrodes' glue
* emergency surgery
* prematurity (born before 37 week PMA)

Max Age: 17 Months | Sex: All
Age Groups: Child
Study Population: Children under 18 months undergoing elective surgery lasting more than 30 minutes.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Cardiac output | Measurements start before the induction of anesthesia and ends at emergence from anesthesia
  Cardiac output will be non-invasivaly measured during the perioperative period by means of electrical electrocardiometry

SECONDARY OUTCOMES:
Association between cardiac output and blood pressure during anesthesia | Time-locked measurements start before the induction of anesthesia and ends at emergence from anesthesia
  Describe how cardiac output and blood pressure are associated in infants during anesthesia
Association between cardiac output and cerebral NIRS during anesthesia | Time-locked measurements start before the induction of anesthesia and ends at emergence from anesthesia
  Describe how cardiac output and cerebral NIRS are associated in infants during anesthesia
Association between cardiac output and other anesthesia factors (concentration of anesthetic agent, carbon dioxide) during anesthesia | Time-locked measurements start before the induction of anesthesia and ends at emergence from anesthesia
  Describe how cardiac output and other anesthesia factors are associated in infants during anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Vutskits, MD PhD, Principal Investigator — University Hosptials of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided